CLINICAL TRIAL: NCT00481416
Title: Evaluation of the PillCam™ Eso Capsule in the Detection of Esophageal Varices
Brief Title: "Evaluation of the PillCam™ESO Capsule in the Detection of Esophageal Varices
Acronym: MA-37
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Collaborators: Ethicon Endo-Surgery (Industry)
Other Study IDs: MA-37
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2006-06

CONDITIONS: Esophageal Varices
Keywords: Esophageal Varices; PillCam Eso; Capsule Endoscopy; Given Imaging; Inscope
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PillCam Eso

SUMMARY:
The purpose of the study is to access the accuracy of the PillCam Eso capsule in identifying the presence of suspected esophageal disease in patients undergoing surveillance or screening for esophageal disease by standard endoscopy

DETAILED DESCRIPTION:
The procedure that is being evaluated in this study is an esophageal capsule which is part of the Given® Diagnostic System. This system has been developed for aiding the gastroenterologist in diagnosing small bowel diseases or disorders, as routine methods used today cannot explore the entire length of the small bowel in detail. It is currently available in more than 50 countries worldwide, including the Europe, USA, Canada, Central and South America, Australia and Asia. More than 300,000 capsules have already been ingested worldwide. In this study, a capsule developed and approved for the esophagus (food tube between the mouth and stomach) with two optical heads (mini cameras) will be used and intended to take better recorded pictures of the esophagus.

During the study the study participant will undergo a capsule endoscopy and an upper esophagoscopy. The method under investigation in this study is the capsule endoscopy.

The capsule endoscope is a small camera, about an inch long and less than half an inch wide, which you will be asked to swallow. The camera travels from a person's mouth all the way through their stomach and intestines and is eventually passed in the stool. The camera has a light source (like a flash on a regular camera) and takes pictures of the esophagus. The pictures are sent to a recorder, about the size of a wallet, using electronic signals for 20 minutes while the wireless endoscope goes through your esophagus. The disposable capsule is passed in the stool in an average of 24 hours.

After the capsule endoscopy the study participant will undergo the esophagoscopy. An esophagoscopy is the standard method used to view the esophagus. It involves inserting a long flexible tube with a light and camera on the end (called an endoscope) through the mouth and down the throat and esophagus. It may also involve the use of a sedative.

The study involves approximately two-three clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has prior endoscopic confirmation of esophageal varices and is undergoing surveillance endoscopy or
2. Patient has sign/symptoms of chronic liver disease, without previous diagnosis of esophageal varices,with clinical indication to undergo esophagoscopy (or EGD)

Exclusion Criteria:

1. Patient has difficulty swallowing
2. Patient has known Zenker's Diverticulum
3. Patient went through previous endoscopic treatment of esophageal varices
4. Patient is known or is suspected to suffer from intestinal obstruction
5. Patient has a cardiac pacemaker or other implanted electro medical device
6. Female patient is pregnant
7. Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule
8. Patient has had a prior abdominal surgery of the gastrointestinal tract (other than uncomplicated appendectomy or uncomplicated cholecystectomy)
9. Patient has any condition, which precludes compliance with study and/or device instructions
10. Patient suffers from life threatening conditions
11. Patient is currently participating in another clinical study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2004-12; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn M Eisen, MD, Principal Investigator — OHSU Portland, OR
Locations (5):
- United States (3):
  - Mayo Clinic Hospital, Scottsdale, Arizona
  - Minnesota Gastroenterology Associates, Plymouth, Minnesota
  - Oregon Health Sciences University, Portland, Oregon
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- See also: Sponsor web site — http://capsuleendoscopy.org